CLINICAL TRIAL: NCT03239587
Title: Investigating the Effect of Simulated Live Piano Music on Preoperative Cancer Patients, Health Care Providers and Hospital Volunteers Using Validated Questionnaires, Proteomic Analysis, and Neuroimaging
Brief Title: Investigating the Effect of Simulated Live Piano Music on Preoperative Cancer Patients, Health Care Providers and Hospital Volunteers Using Validated Questionnaires and Proteomic Analysis
Status: Withdrawn | Type: Observational
Why Stopped: No participants
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-0808
Record Dates: First submitted 2017-08-02; First posted 2017-08-04 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Symptoms and Signs Involving Cognition Perception Emotion & Behaviour; Abdominal Cancer Patients
Keywords: Symptoms and signs involving cognition perception emotion & behaviour; Abdominal cancer patients; Musical preop intervention; Surveys; Questionnaires; Blood draws
MeSH Terms: conditions — Behavior | interventions — Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood (about 1½ teaspoons each time) drawn before and about 30 minutes after participant either listens to music or stands in the waiting room without music.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No Musical Intervention - Control Group: Participants wait for 30 minutes in a standard pre-surgery waiting area without music.
  Blood drawn before, and about 30 minutes after participant stands in the waiting room without music.
  Participants complete 2 questionnaires about anxiety and stress levels.
  Interventions: Procedure: Blood Draws; Behavioral: Questionnaires
- Musical Intervention Group: Participants wait for 30 minutes in waiting area with a Steinway Spirio grand piano that plays 30 minutes of simulated piano music.
  Blood drawn before, and about 30 minutes after participant in the waiting room with a Steinway Spirio grand piano that plays 30 minutes of simulated piano music.
  Participants complete 2 questionnaires about anxiety and stress levels.
  Interventions: Behavioral: Musical Intervention; Procedure: Blood Draws; Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Musical Intervention — Participants wait for 30 minutes in waiting area with a Steinway Spirio grand piano that plays 30 minutes of simulated piano music.
  Groups: Musical Intervention Group
Procedure: Blood Draws — No Musical Intervention - Control Group: Blood drawn before, and about 30 minutes after participant stands in the waiting room without music.
  Musical Intervention Group: Blood drawn before, and about 30 minutes after in waiting room with a Steinway Spirio grand piano that plays 30 minutes of simulated piano music.
Behavioral: Questionnaires — Participants complete 2 questionnaires about anxiety and stress levels. It should take about 20-30 minutes to complete.
  Other Names: Surveys

SUMMARY:
The goal of this research study is to learn if simulated live piano music can change the amount of stress felt in patients with cancer before surgery, health care providers caring for cancer patients, and/or hospital volunteers.

This is an investigational study.

Up to 304 participants (200 patients, 52 volunteers, and 52 healthcare providers) will be enrolled in this study. All will take part at MD Anderson.

DETAILED DESCRIPTION:
If you agree to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups. Participants in the first group will wait for 30 minutes in a standard pre-surgery waiting area without music. Participants in the other group will go to a waiting room with a Steinway Spirio grand piano that plays 30 minutes of simulated piano music.

A Steinway Spirio grand piano is a special type of piano that plays music by itself (also called a player piano). The music will be chosen by the study staff and pre-recorded on the piano. Although the keys will move on the piano as if someone is playing the piano, you will be alone in the room.

You will have an equal chance (50/50) of being assigned to either group. Both you and the person in charge of this study will know to which group you have been assigned. You do not get to choose which group you are in.

Study Procedures:

Before and about 30 minutes after you either listen to music or stand in the waiting room without music:

* Blood (about 1½ teaspoons each time) will be drawn to learn how your body is responding to the music or silence by measuring the amount of cortisol in your body (a type of hormone related to stress) and for biomarker testing. Biomarkers are found in the blood and may be related to your reaction to the music or silence. If you are a healthcare provider or volunteer, you will not have these blood draws.
* You will complete 2 questionnaires about your anxiety and stress levels. It should take about 20-30 minutes to complete.

Length of Study:

You participation on this study will be over after the last blood draw and questionnaire are completed.

ELIGIBILITY:
Inclusion Criteria:

1) Patients: To preserve a homogenous cohort and comply with the departmentally-organized research infrastructure, we will include pPreoperative abdominal cancer patients undergoing surgery, or healthcare provider from all specialties at MDACC or volunteer from MDACC Volunteer Service.

Exclusion Criteria:

1. Cannot give informed consent
2. Are deaf or hearing-disabled
3. Less than 18 years in age
4. Profess extreme dislike of music.
5. Wait time is longer than 240 min.
6. Underlying structural brain abnormality or neurologic comorbidity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer participants waiting for surgery at UT MD Anderson Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2018-04-24 (Actual); Study Completion 2018-04-24 (Actual)

PRIMARY OUTCOMES:
Effect of Defined Musical Intervention on Perceived Stress in Preoperative Cancer Participants | 1 day
  Effect of defined musical intervention on perceived stress measured by the Spielberger State-Trait Anxiety Inventory (STAI-S).

CONTACTS AND LOCATIONS:
Overall Officials: Claudius Conrad, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org